CLINICAL TRIAL: NCT00496678
Title: RCT of Primary Care-based Patient Navigation-Activation
Brief Title: Trial of Patient Navigation-Activation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Kevin Fiscella M.D. MPH, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RO1U01CA116924
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2007-12

CONDITIONS: Breast Cancer; Colorectal Cancer
Keywords: PNRP; navigation; navigator; activation; disparities; randomized control trial; primary care; racial and ethnic minorities
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navigation (Experimental): Navigation through the cancer care system is the intervention
  Interventions: Behavioral: Navigation
- Standard of Care (Active Comparator): Cancer patient receives standard of care.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Navigation — Cancer patients are randomly assigned to receive standard of care or the help of a trained person to navigated them through the cancer care system
  Arms: Navigation
Behavioral: Standard of Care — Cancer patients receive standard of care for their cancer treatment
  Arms: Standard of Care

SUMMARY:
The University of Rochester, Department of Family Medicine, funded by the National Cancer Institute will train community health workers to guide patients through the cancer care system. The project will help to teach patients how to communicate more effectively with their health care team in order to understand the treatment options available to them. Although not widely available, it is believed patient navigation programs are beneficial.

This research study will evaluate how well this tool works, especially among those who experience disparities in health care. The goal is to determine if having a trained navigator shortens the time between an abnormal test result and a definitive diagnosis and between a definitive diagnosis and completion of treatment for breast and colorectal cancer patients. The project also will evaluate whether navigation improves the ability to communicate with the doctor, patient satisfaction with care and quality of life.

DETAILED DESCRIPTION:
Racial and ethnic minority groups and low-income persons experience significantly higher cancer mortality rates than other Americans. These disparities are due to at least two factors: (1) delays in follow-up of abnormal cancer screening results and (2) suboptimal management of diagnosed cancer. Patient navigation represents a promising means for addressing disparities by improving cancer related management for minority and other underserved populations. However, patient navigation for cancer has yet to be evaluated through a well-designed randomized controlled trial. Furthermore, patient navigation is likely to prove most effective and sustainable when it is integrated into primary care and helps patients be more active in their care. This combination of patient empowerment and enablement is referred to as "activation." The aim of this project is to evaluate the effectiveness and costs of such a program in a rigorous manner so that the results can be generalized and the program can be widely disseminated and implemented. we will develop, implement, and evaluate a primary care-based, patient navigation-activation program using specially-trained community health workers (CHWs). We propose to investigate the effect of this intervention on timing and quality of cancer-related care. Secondary aims examine the impact of navigation on disparities in care, improvement in patient activation and total costs. Project findings will inform national policy regarding patient navigation for cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Receive care at a participating practice
2. Have received a positive breast or colorectal cancer screening test requiring follow-up on a different day
3. Have been newly diagnosed with breast or colorectal cancer
4. Have received notification by the provider of an abnormal breast or colorectal screening result

Exclusion Criteria:

1. Cognitively impaired
2. Institutionalized (nursing home, incarcerated)
3. Children <18
4. Actively involved in cancer treatment at time of presentation
5. Currently or previously navigated with (a) navigation documented in the medical record or (b) patient can articulate that they are in a navigation program or case management program for cancer
6. History of prior invasive cancer, lymphoma, or leukemia except non-melanoma (basal or squamous of the skin) cancer or CIN (Cervical intraepithelial neoplasia).
7. Prior cancer that has been treated-The rationale for excluding patients with any prior cancers that have been treated is that patient familiarity with the treatment process in general would make care easier even without a navigator.
8. Women who are pregnant at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To develop, implement, and evaluate a primary care-based, patient navigation program using specially-trained community health workers. We will investigate the effect of this intervention on timing and quality of cancer-related care. | 5 years

SECONDARY OUTCOMES:
Secondary aims examine the impact of navigation on disparities in care, improvement in patient activation and total costs. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fiscella, M.D., MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Battaglia TA, Darnell JS, Ko N, Snyder F, Paskett ED, Wells KJ, Whitley EM, Griggs JJ, Karnad A, Young H, Warren-Mears V, Simon MA, Calhoun E. The impact of patient navigation on the delivery of diagnostic breast cancer care in the National Patient Navigation Research Program: a prospective meta-analysis. Breast Cancer Res Treat. 2016 Aug;158(3):523-34. doi: 10.1007/s10549-016-3887-8. Epub 2016 Jul 18. PMID 27432417
- [Derived] Wells KJ, Winters PC, Jean-Pierre P, Warren-Mears V, Post D, Van Duyn MA, Fiscella K, Darnell J, Freund KM; Patient Navigation Research Program Investigators. Effect of patient navigation on satisfaction with cancer-related care. Support Care Cancer. 2016 Apr;24(4):1729-53. doi: 10.1007/s00520-015-2946-8. Epub 2015 Oct 5. PMID 26438146
- [Derived] Rodday AM, Parsons SK, Snyder F, Simon MA, Llanos AA, Warren-Mears V, Dudley D, Lee JH, Patierno SR, Markossian TW, Sanders M, Whitley EM, Freund KM. Impact of patient navigation in eliminating economic disparities in cancer care. Cancer. 2015 Nov 15;121(22):4025-34. doi: 10.1002/cncr.29612. Epub 2015 Sep 8. PMID 26348120
- [Derived] Ko NY, Darnell JS, Calhoun E, Freund KM, Wells KJ, Shapiro CL, Dudley DJ, Patierno SR, Fiscella K, Raich P, Battaglia TA. Can patient navigation improve receipt of recommended breast cancer care? Evidence from the National Patient Navigation Research Program. J Clin Oncol. 2014 Sep 1;32(25):2758-64. doi: 10.1200/JCO.2013.53.6037. Epub 2014 Jul 28. PMID 25071111
- [Derived] Hendren S, Griggs JJ, Epstein RM, Humiston S, Rousseau S, Jean-Pierre P, Carroll J, Yosha AM, Loader S, Fiscella K. Study protocol: a randomized controlled trial of patient navigation-activation to reduce cancer health disparities. BMC Cancer. 2010 Oct 13;10:551. doi: 10.1186/1471-2407-10-551. PMID 20939928